CLINICAL TRIAL: NCT05480137
Title: The Efficacy of Scoring Balloon Angioplasty in the Treatment of Chronic Thromboembolic Pulmonary Hypertension Based on Optical Coherence Tomography：A Single-center Randomized Controlled
Brief Title: OCT Evaluates the Effects of CTEPH Treated by Scoring Balloon
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Wei Huang, Professor, First Affiliated Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022XMSB0000725
Record Dates: First submitted 2022-07-25; First posted 2022-07-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: CTEPH

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- plain balloon (Other): plain balloon is used in BPA
  Interventions: Procedure: NSE scoring balloon and plain balloon angioplasty
- NSE scoring balloon (Other): NSE scoring balloon is used in BPA
  Interventions: Procedure: NSE scoring balloon and plain balloon angioplasty

INTERVENTIONS:
Procedure: NSE scoring balloon and plain balloon angioplasty — Using NSE scoring balloon or plain balloon in BPA surgery.

SUMMARY:
Chronic thromboembolic pulmonary hypertension (CTEPH) is a disease of obstructive pulmonary artery remodelling as a consequence of major vessel thromboembolism.

The diagnosis of CTEPH is based on findings obtained after at least 3 months of effective anticoagulation in order to discriminate this condition from subacute PE. These findings are mean pulmonary artery pressure ≥25mmHg with pulmonary artery wedge pressure ≤15 mmHg, mismatched perfusion defects on lung scan and specific diagnostic signs for CTEPH seen by multidetector CT angiography, MR imaging or conventional pulmonary cineangiography, such as ring-like stenoses, webs/slits and chronic total occlusions (pouch lesions or tapered lesions). Balloon pulmonary angioplasty (BPA) is a type of effective treatment for CTEPH. Plain balloon is usually used in BPA surgery,however，the efficacy and safety of NSE scoring balloon in BPA is not clear. Optical coherence tomography（OCT）as a good assessment methods has been reported. Our study aims to explore the efficacy and safty of NSE scoring balloon based on OCT in BPA .

DETAILED DESCRIPTION:
After right heart catheterization,BPA procedures are performed via femoral vein approach. 8-Fr sheath is inserted into the vein and 6-Fr guiding cathater was advanced to the main pulmonary artery through the 8-Fr guiding catheter using a 0.035-inch wire. We select a branch of the pulmonary artery by a 6-Fr guiding catheter (JR4.0). Pulmonary angiography is performed manually using half contrast medium diluted with saline. A 0.014-inch guidewire (Sion) is crossed under the pulmonary angiography, and OCT (Fig.1: Types of lesions) is used for the detection of Lumen diameter (mm), Intimal thickness (mm), Intimal area (mm2), Intimal thickness/lumen diameter, Intimal area/lumen area, which are defined as short diameter assessed by OCT. The balloon size, the expansion pressure and the choice of scoring balloon or plain balloon angioplasty are at the discretion of the operator. Balloon-to-vessel (B/V) ratio is defined as the balloon diameter divided by vessel diameter assessed with OCT (1:0.7-1). Pulmonary arteries with an inner diameter of less than 4mm detected by OCT were selected for BPA performance. Scoring balloon and plain balloon are used in half of pulmonary lesions respectively., use the Plain balloon was used to predilate, If the vascular Lesion is a completely occlusive or the scoring balloon cannot pass through vessels.

ELIGIBILITY:
Inclusion Criteria:

1. PEA not available in patients with CTEPH
2. Patients assessed by a multidisciplinary panel as having a large risk-benefit ratio for PEA surgery
3. Patients with postoperative residual pulmonary hypertension after PEA
4. Patients with CTEPH not respond well to medical treatment

Exclusion Criteria:

1. Other cardiovascular diseases, such as Congenital heart disease, valvular disease, cardiomyopathy, aortic dissection, arteritis, arrhythmia, Severe heart failure
2. Other diseases of the respiratory system, such as chronic obstructive pulmonary disease, asthma, pulmonary bronchial artery embolism, and other diseases, such as vasculitis, Pulmonary sarcoma, etc.
3. central-type chronic thromboembolic pulmonary hypertension
4. Other types of PAH except CTEPH
5. malignant tumor patients
6. severe renal dysfunction （GFR <30ml/min）
7. iodine contrast medium allergy
8. Gravida
9. high risk of serious bleeding：Active bleeding，Acute stroke，Severe hepatic insufficiency (Child-Pugh C)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2020-08-30 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
PVR after BPA | 1-3 months after BPA
  Mean pulmonary artery pressure (mPAP), mean pulmonary wedge pressure (mPCWP) and cardiac output （CO） will be combined to report pulmonary vascular resistance (PVR）in Unit Wood. Formula： PVR=（mPAP-mPCWP）/CO

CONTACTS AND LOCATIONS:
Overall Officials: Rui Xiang, Phd, Study Chair — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- the First Affiliated Hospital, Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
All IPD will be shared with other researchers
Time Frame: After our study is published
Access Criteria: IPD shares with experienced and high-volume CTEPH centres.